CLINICAL TRIAL: NCT01831193
Title: Effect of Oral Supplementation With Curcumin (Turmeric) in Patients With Proteinuric Chronic Kidney Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Instituto Nacional de Cardiologia Ignacio Chavez (Other)
Responsible Party: Principal Investigator, Magdalena Madero, MD, Instituto Nacional de Cardiologia Ignacio Chavez
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 12-793
Record Dates: First submitted 2013-04-09; First posted 2013-04-15 (Estimated); Last update posted 2014-07-24 (Estimated); Status verified 2014-07

CONDITIONS: Proteinuria
MeSH Terms: conditions — Proteinuria | interventions — Curcumin

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Diabetic (Active Comparator)
  Interventions: Drug: Curcumin
- Non-diabetic (Active Comparator)
  Interventions: Drug: Curcumin

INTERVENTIONS:
Drug: Curcumin
  Other Names: Turmeric

SUMMARY:
The purpose of this study is to determine if the oral supplementation with curcumin reduces proteinuria in patients with chronic kidney disease regardless the ethiology.

DETAILED DESCRIPTION:
Curcumin is a potent antioxidant found in extracts of the rhizome of the plant Curcuma longa L.

Different studies have demonstrated that curcumin has potent biological activity and therefore is an effective therapeutic agent for the treatment of various ailments.

This compound acts as a bifunctional antioxidant:

ه is capable of reacting directly with highly reactive oxygen species. ه acts indirectly by its ability to induce the expression of various cytoprotective proteins through Keap1/Nrf2/ARE pathway.

Although RAAS blockade is the cornerstone to prevent the progression of proteinuric nephropathy, a significant number of patients remained with proteinuria and progress to end-stage renal disease.

Due to the low cost and few side effects of curcumin, this could become an adjuvant treatment of proteinuric nephropathy purposes attenuate the progression of chronic kidney disease.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of proteinuric chronic kidney disease with 1g or more of proteins in a daily recollection.
* Individuals taking Angiotensin II Receptor Blocker or ACE inhibitors in monotherapy with maximum dose or in combination.

Exclusion Criteria:

* Hepatic damage.
* Malignancy.
* Pregnancy.
* Peritoneal or hemodialysis.
* Organ transplantation.
* Heart failure classification III or IV (New York Heart Association).
* History of chemotherapy within 2 years prior to screening.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2013-02; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Change in proteinuria | 8 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto Nacional de Cardiologia Ignacio Chavez, Mexico City, Mexico City, Mexico

REFERENCES:
- [Derived] Colombijn JM, Hooft L, Jun M, Webster AC, Bots ML, Verhaar MC, Vernooij RW. Antioxidants for adults with chronic kidney disease. Cochrane Database Syst Rev. 2023 Nov 2;11(11):CD008176. doi: 10.1002/14651858.CD008176.pub3. PMID 37916745